CLINICAL TRIAL: NCT03455738
Title: Dynamic Arterial Elastance Measured by Uncalibrated Pulse Contour Analysis Predicts Arterial Pressure Response to a Decrease in Norepinephrine (VESA) Dynamic Arterial Elastance Measured by Uncalibrated Pulse Contour Analysis
Brief Title: Dynamic Arterial Elastance Measured by Uncalibrated Pulse Contour Analysis Predicts Arterial Pressure Response to a Decrease in Norepinephrine
Acronym: VESA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-28
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Vasoplegia Syndrome
Keywords: Vasoplegia, norepinephrine, dynamic arterial elastance
MeSH Terms: conditions — Vasoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: vasoplegic syndrome — Patients with vasoplegic syndrome for whom the intensive care physician planned to decrease the norepinephrine dosage were included. Hemodynamic and uncalibrated pulse contour analysis (Volume view, FloTrac, Edwards Lifescience, Irvine) values were obtained before and after decreasing the norepineprhine dosage. Responders were defined by a >10% decrease in mean arterial pressure (MAP).

SUMMARY:
Dynamic arterial elastance (Eadyn) has been proposed as an indicator of arterial tone that can predict norepinephrine-dependent arterial pressure. Eadyn is calculated using the ratio of respiratory pulse pressure variation (PPV) over the respiratory stroke volume variation (SVV). Guinot et al demonstrated a decrease in the duration of norepinephrine treatment with the use of Eadyn. To date, studies that have validated Eadyn at bedside have used cardiac output (CO) calibrated pulse contour analysis (PiCCO™, Pulsion™) or oesophageal doppler. Such monitoring systems need dedicated and specific arterial line and venous access that may limit their use at bedside. In addition to CO calibrated pulse contour analysis, CO uncalibrated pulse contour analysis has been developed and is considered less invasive. Nevertheless, one limitation of the latter CO monitoring is inaccuracy of CO measurement in patients who are being treated with norepinephrine. These limitations may affect the predictability of Eadyn. We conducted a prospective study in a university hospital ICU. Patients with vasoplegic syndrome for whom the intensive care physician planned to decrease the norepinephrine dosage were included. Hemodynamic and uncalibrated pulse contour analysis (Volume view, FloTrac, Edwards Lifescience, Irvine) values were obtained before and after decreasing the norepinephrine dosage. Responders were defined by a >10% decrease in mean arterial pressure (MAP).

DETAILED DESCRIPTION:
* Background : Dynamic arterial elastance (Eadyn) has been proposed as an indicator of arterial tone that can predict norepinephrine-dependent arterial pressure. Eadyn is calculated using the ratio of respiratory pulse pressure variation (PPV) over the respiratory stroke volume variation (SVV). Guinot et al demonstrated a decrease in the duration of norepinephrine treatment with the use of Eadyn. To date, studies that have validated Eadyn at bedside have used cardiac output (CO) calibrated pulse contour analysis (PiCCO™, Pulsion™) or oesophageal doppler. Such monitoring systems need dedicated and specific arterial line and venous access that may limit their use at bedside. In addition to CO calibrated pulse contour analysis, CO uncalibrated pulse contour analysis has been developed and is considered less invasive. Nevertheless, one limitation of the latter CO monitoring is inaccuracy of CO measurement in patients who are being treated with norepinephrine. These limitations may affect the predictability of Eadyn.
* Purpose : To date, no study has evaluated the ability of Eadyn measured by uncalibrated pulse contour analysis to assess arterial pressure response to a decreased dose of norepinephrine. We tested the hypothesis that Eadyn calculated from uncalibrated pulse contour analysis predicts the arterial-pressure response to a norepinephrine decrease in patients treated with norepinephrine

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were all consecutive patients with a diagnosis of vasoplegic syndrome, treated with norepinephrine, for whom the attending physician decided to decrease the norepinephrine dosage. The vasoplegic syndrome was defined as persistent arterial hypotension with normal or high cardiac output and low systemic vascular resistance

Exclusion Criteria:

Exclusion criteria were patients treated with epinephrine and/or dobutamine, arrhythmia, intra-abdominal hypertension and patients younger than 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: one group Patients with vasoplegic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Dynamic arterial elastance (Eadyn) defined as the ratio of PPV/SVV calculated from uncalibrated pulse contour analysis | 60 minutes